CLINICAL TRIAL: NCT05466396
Title: Lung Health of Early Chronic Obstructive Pulmonary Disease: A Multi-center Cohort Study
Brief Title: Lung Health of Early COPD: A Multi-center Cohort Study
Acronym: LHEC
Status: Recruiting | Type: Observational
Sponsor: Ting YANG (Other)
Collaborators: Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, Ting YANG, Vice Director of Respiratory Center, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Other Study IDs: LHEC
Record Dates: First submitted 2022-07-17; First posted 2022-07-20 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: COPD
Keywords: early COPD; spirometry; lung health
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Smoking Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine and sputum simple will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Smokers with Pre-COPD: Smoking history ≥ 10 pack-years 0.7≤ FEV1/FVC<0.8 and FEV1%pred ≥ 80% (post-bronchodilator)
  Interventions: Behavioral: smoking
- Smokers with Mild-COPD: Smoking history ≥ 10 pack-years FEV1/FVC<0.7 and FEV1%pred ≥ 80% (post-bronchodilator)
  Interventions: Behavioral: smoking
- Non-Smokers with Pre-COPD: Smoking history < 10 pack-years or never-smokers 0.7≤ FEV1/FVC<0.8 and FEV1%pred ≥ 80% (post-bronchodilator)
- Non-Smokers with Mild-COPD: Smoking history < 10 pack-years or never-smokers FEV1/FVC<0.7 and FEV1%pred ≥ 80% (post-bronchodilator)
- Healthy Controls: Healthy volunteers without smoking history FEV1/FVC ≥ 0.8 and FEV1%pred ≥ 80% (post-bronchodilator)

INTERVENTIONS:
Behavioral: smoking — Smoking history and spirometry are used to define groups
  Groups: Smokers with Mild-COPD; Smokers with Pre-COPD

SUMMARY:
This is a multi-center, prospective, cohort study in early COPD patients. This study aims to elucidate the lung function decline and its association with smoking and other risk factors. Other biomarkers and image markers from chest CT scan are also analyzed to investigate the lung function in early COPD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Gender: male or female
2. Age: 35-75 years old
3. post-bronchodilator spirometry: FEV1/FVC < 0.8 and FEV1%pred ≥80%

Exclusion Criteria:

1. Other diseases may affect lung function, like lung cancer, bronchiectasis, interstitial lung disease or chest surgery.
2. BMI > 35 kg/m2
3. Dementia or other severe neurological disease
4. Pregnancy
5. Conditions that contraindicated lung function test

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers with mild lung function abnormality will be included in this cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 1550 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Lung function decline in Pre-COPD and Mild-COPD patients | 2 years
  FEV1 decline in Pre-COPD and Mild-COPD patients

SECONDARY OUTCOMES:
Lung function decline in smokers with Pre-COPD and Mild-COPD | 2 years
  FEV1 decline in smokers with Pre-COPD and Mild-COPD
Lung function decline in non-smokers with Pre-COPD and Mild-COPD | 2 years
  FEV1 decline in non-smokers with Pre-COPD and Mild-COPD

OTHER OUTCOMES:
Lung function decline and biomarkers in Pre-COPD and Mild-COPD patients | 2 years
  Association between FEV1 decline and biomarkers in blood, sputum or urine in Pre-COPD and Mild-COPD patients
Lung function decline and Image markers in Pre-COPD and Mild-COPD patients | 2 years
  Association between FEV1 decline and structural markers form chest CT scan in Pre-COPD and Mild-COPD patients

CONTACTS AND LOCATIONS:
Overall Officials: Ting Yang, M.D., Principal Investigator — China-Japan Friendship Hospital
Locations (2):
- China (2):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li W, Lei J, Li B, Tang X, Peng Y, Huang K, Yang T. Lung Health of Early COPD (LHEC): A Multi-Center Cohort Study-Rational and Design. Int J Chron Obstruct Pulmon Dis. 2025 Jul 19;20:2561-2568. doi: 10.2147/COPD.S517185. eCollection 2025. PMID 40703223